CLINICAL TRIAL: NCT06636851
Title: Effect of Site of Right Ventricular (RV) Pacing on RV Function, Left Ventricular (LV) Dyssynchrony and Contraction Efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mustafa Mohamed Ahmed Mohamed Ali, Dr, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RV Pacemaker lead location
Record Dates: First submitted 2024-09-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Heart Block; Heart Block Complete; Systolic Function
Keywords: pacemaker; RV function; LV function; GLS
MeSH Terms: conditions — Heart Block | interventions — Defibrillators

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RV Apical pacing (Active Comparator): Patient with the pacemaker RV lead located at the RV apex
  Interventions: Device: Pacemaker and defibrillator
- RV Septal pacing (Active Comparator): Patient with the pacemaker RV lead located at the RV septum.
  Interventions: Device: Pacemaker and defibrillator

INTERVENTIONS:
Device: Pacemaker and defibrillator — Permenant pacemaker implantation with lead fixed to the RV Septal location
  Other Names: Pacemaker lead location to the RV septum
  Arms: RV Septal pacing
Device: Pacemaker and defibrillator — Description: Permenant pacemaker implantation with lead fixed to the RV Apical location
  Other Names: Pacemaker lead location to the RV Apex
  Arms: RV Apical pacing

SUMMARY:
To evaluate RV systolic function and LV mechanical dyssynchrony and function in different lead position in the RV during permanent pacemaker implantation by using speckle tracking echocardiography (STE) and 3D volumetric ejection fraction

DETAILED DESCRIPTION:
Permanent pacing with right ventricular stimulation is the standard method used in patients with bradyarrhythmia, and recommended by current international guidelines because it is associated with improved clinical outcomes. The extent of right ventricular pacing (RVP) varies between patients and many individuals tolerate a high proportion of RVP without complications. However, chronic RVP may cause electrical and mechanical dyssynchrony that may lead to impaired left ventricular ejection fraction (LVEF). Dyssynchronous ventricles require more oxygen to generate the same amount of mechanical work and the consequence is a decline in the efficieny of myocardial contraction. RV septal pacing (RVS) is thought to allow more physiological LV depolarisation, than RV apical pacing (RVA) with preservation of LV function. However, there are conflicting data on its benefits, and the recently completed Protect-Pace (The protection of LV function during RV pacing) study showed both RVA and non-RVA pacing to have a small adverse effect on EF in patients with preserved LV function, but no difference between the methods. The effect of RV pacing on RV function has not been evaluated systematically, with most studies focusing on tricuspid regurgitation (TR) as the outcome of interest. Echocardiographic assessment of LV dyssynchrony has been extensively used because it is noninvasive, widely available, and has no known risk or side effect. Speckle tracking echocardiography is a novel echocardiographic technique without the angle dependence of an ultrasound beam and is able to measure regional deformation in any direction in the LV and RV, that can detect subtle myocardial dysfunction because it is more sensitive compared with conventional parameters, Furthermore, strain imaging can display the timing and extent of myocardial thickening and stretching so that it is well suited to estimate the amount of inefficient dyssynchronous contraction. Global Longitudinal Strain (GLS) and LV mechanical function and dyssynchrony assessment by speckle-tracking echocardiography (STE) enables us to detect subclinical LV dysfunction. And also a very attractive clinical tool for the assessment of right ventricular (RV) systolic performance, providing incremental diagnostic and prognostic information over the traditional indices of RV function, Among various imaging modalities, echocardiography is currently the method of choice for clinical assessment of RV longitudinal strain (RVLS). The methodology of speckle-tracking echocardiography to obtain RVLS has been recently standardized and demonstrated to be feasible, accurate, and robust for clinical use. Inter-technique and inter-vendor comparability and reliability of RVLS are improving. RVLS is advantageous because it is more sensitive to subtle changes in myocardial function than conventional parameters used to assess RV function (i.e. tricuspid annular plane systolic excursion, tissue Doppler systolic velocity, fractional area change, or RV ejection fraction) representing a sensitive tool for the long-term follow-up of patients.

ELIGIBILITY:
Inclusion Criteria:

- Patients with symptomatic bradycardia indicated for permanent pacemaker implantation according to recent European guidelines.

Exclusion Criteria:

* Patients with reduced RV function.
* Patients with reduced LV systolic function.
* Significant valvular lesions.
* Congenital heart disease that might affect RV and/or LV function.
* Patients undergoing CRT or Implantable Cardioverter-Defibrillator (ICD).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
To detect a 3% difference in Longitudinal Strain (GLS) between groups. | 6 months
  To detect a 3% difference in Longitudinal Strain (GLS) between group A (right ventricular apex) and the group B (right ventricular septum).
  A standard deviation of 4% was used for the sample size calculation based on previous studies

CONTACTS AND LOCATIONS:
Overall Officials: Minia University, Study Director — Minia University, faculty of medicine
Locations (1):
- South Valley University, Qena Governorate, Qena Governorate, Egypt

REFERENCES:
- [Background] Saito M, Iannaccone A, Kaye G, Negishi K, Kosmala W, Marwick TH; PROTECT-PACE investigators. Effect of Right Ventricular Pacing on Right Ventricular Mechanics and Tricuspid Regurgitation in Patients With High-Grade Atrioventricular Block and Sinus Rhythm (from the Protection of Left Ventricular Function During Right Ventricular Pacing Study). Am J Cardiol. 2015 Dec 15;116(12):1875-82. doi: 10.1016/j.amjcard.2015.09.041. Epub 2015 Oct 9. PMID 26517949
- [Background] Michalik J, Dabrowska-Kugacka A, Kosmalska K, Moroz R, Kot A, Lewicka E, Szolkiewicz M. Hemodynamic Effects of Permanent His Bundle Pacing Compared to Right Ventricular Pacing Assessed by Two-Dimensional Speckle-Tracking Echocardiography. Int J Environ Res Public Health. 2021 Nov 8;18(21):11721. doi: 10.3390/ijerph182111721. PMID 34770235
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy: Developed by the Task Force on cardiac pacing and cardiac resynchronization therapy of the European Society of Cardiology (ESC) With the special contribution of the European Heart Rhythm Association (EHRA). Rev Esp Cardiol (Engl Ed). 2022 May;75(5):430. doi: 10.1016/j.rec.2022.04.004. No abstract available. English, Spanish. PMID 35525571
- [Background] Van De Heyning CM, Elbarasi E, Masiero S, Brambatti M, Ghazal S, Al-Maashani S, Capucci A, Leong D, Shivalkar B, Saenen JB, Miljoen HP, Morillo CA, Divarakarmenon S, Amit G, Ribas S, Baiocco E, Maolo A, Romandini A, Maffei S, Connolly SJ, Healey JS, Dokainish H. Prospective Study of Tricuspid Regurgitation Associated With Permanent Leads After Cardiac Rhythm Device Implantation. Can J Cardiol. 2019 Apr;35(4):389-395. doi: 10.1016/j.cjca.2018.11.014. Epub 2018 Nov 29. PMID 30852048
- [Background] Kaye GC, Linker NJ, Marwick TH, Pollock L, Graham L, Pouliot E, Poloniecki J, Gammage M; Protect-Pace trial investigators. Effect of right ventricular pacing lead site on left ventricular function in patients with high-grade atrioventricular block: results of the Protect-Pace study. Eur Heart J. 2015 Apr 7;36(14):856-62. doi: 10.1093/eurheartj/ehu304. Epub 2014 Sep 4. PMID 25189602
- [Background] Khurshid S, Epstein AE, Verdino RJ, Lin D, Goldberg LR, Marchlinski FE, Frankel DS. Incidence and predictors of right ventricular pacing-induced cardiomyopathy. Heart Rhythm. 2014 Sep;11(9):1619-25. doi: 10.1016/j.hrthm.2014.05.040. Epub 2014 Jun 2. PMID 24893122
- [Background] Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, Cleland J, Deharo JC, Delgado V, Elliott PM, Gorenek B, Israel CW, Leclercq C, Linde C, Mont L, Padeletti L, Sutton R, Vardas PE; ESC Committee for Practice Guidelines (CPG); Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Kirchhof P, Blomstrom-Lundqvist C, Badano LP, Aliyev F, Bansch D, Baumgartner H, Bsata W, Buser P, Charron P, Daubert JC, Dobreanu D, Faerestrand S, Hasdai D, Hoes AW, Le Heuzey JY, Mavrakis H, McDonagh T, Merino JL, Nawar MM, Nielsen JC, Pieske B, Poposka L, Ruschitzka F, Tendera M, Van Gelder IC, Wilson CM. 2013 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy: the Task Force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Eur Heart J. 2013 Aug;34(29):2281-329. doi: 10.1093/eurheartj/eht150. Epub 2013 Jun 24. No abstract available. PMID 23801822
- [Background] Candan O, Gecmen C, Bayam E, Guner A, Celik M, Dogan C. Mechanical dispersion and global longitudinal strain by speckle tracking echocardiography: Predictors of appropriate implantable cardioverter defibrillator therapy in hypertrophic cardiomyopathy. Echocardiography. 2017 Jun;34(6):835-842. doi: 10.1111/echo.13547. Epub 2017 Apr 26. PMID 28444773
- [Background] Abdin A, Yalin K, Zink MD, Napp A, Gramlich M, Marx N, Schuett K. Incidence and predictors of pacemaker induced cardiomyopathy: A single-center experience. J Electrocardiol. 2019 Nov-Dec;57:31-34. doi: 10.1016/j.jelectrocard.2019.08.016. Epub 2019 Aug 23. PMID 31473477